CLINICAL TRIAL: NCT03134924
Title: Vaginal Practices in Human Immunodeficiency Virus (HIV) Positive Women in Zambia, a Bio-Behavioral Intervention "WASH-2"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Maria Alcaide, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120418
Record Dates: First submitted 2017-04-21; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Vaginosis, Bacterial
Keywords: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Sexual Health; Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: The interventional study model used a parallel design, where an enhanced standard of care and intervention were used.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study statistician did not participate in randomization and the recruiter and laboratory personnel were blinded to the condition assignment. The participant was blind to their condition assignment. The reading of all the slides used to diagnose BV was performed by one trained laboratory technician blinded to the participant condition assignment. In case of unclear reading, the slide was reviewed by a second technician and the chief of the laboratory until an agreement was achieved; both the second technician and the chief of the laboratory were blind to the condition assignment of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition (Experimental): The WASH (Women's and Sexual Health) intervention included the elements of the enhanced standard of care condition and in addition, a group-based, culturally-tailored intervention to enhance the uptake of the recommendations. Facilitators covered an intervention manual on risks associated with IVP, symptoms of vaginal infections, vaginal health, women's experience with alternative methods for vaginal care, and communication with partners about vaginal health and the risks associated with IVP.
  Interventions: Behavioral: Women's and Sexual Health [WASH]
- Enhanced Standard of Care (Other): This study provided an "enhanced standard of care" (SOC+) comparison condition, consisting of a genital tract examination, collection of a vaginal swab with gram stain of vaginal secretions, diagnosis of BV using the Nugent criteria and provision of medication (oral metronidazole) within 48 hours of the examination in women with Nugent score of 7-10, regardless of the presence of symptoms. In addition, at baseline, participants received an individual education session on the risk of engaging in IVP, advice to discontinue IVP, and tips for healthy vaginal hygiene, emphasizing avoiding IVP and suggesting replacing IVP by external vaginal cleansing.
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Women's and Sexual Health [WASH] — The WASH was a group-based, 45-minute group session on vaginal health and healthy vaginal practices led by two trained facilitators. The sessions covered topics related to vaginal practices and the potential harm of vaginal practices.
  Other Names: WASH
  Arms: Experimental condition
Behavioral: Enhanced Standard of Care — The "enhanced standard of care" (SOC+) condition received a genital tract examination, collection of a vaginal swab with gram stain of vaginal secretions, diagnosis of BV, and medication as needed. At baseline participants received an individual education session on the risk of engaging in IVP and tips on discontinuing IVP.
  Arms: Enhanced Standard of Care

SUMMARY:
Intravaginal practices (IVP) (cleansing or introducing products inside the vagina for hygiene, health or to please sexual partners) are common among women with HIV. IVP increase the risk of developing bacterial Vaginosis (BV), the most common genital infection associated with transmission of sexually transmitted infections and HIV. This study tested a pilot intervention to reduce IVP and BV in HIV infected women in Zambia. A total of 128 HIV infected women engaging in IVP were randomized to two conditions: enhanced standard of care (n = 70) and experimental (n = 58). All participants received a brief educational counseling session on discontinuation of IVP, and those with BV, were provided with medical treatment for BV. Women in the experimental condition received an additional group-based, culturally tailored intervention. Participants completed questionnaires assessing sexual risk factors and IVP and were assessed for BV using Nugent criteria at baseline, 6 months and 12 months.

DETAILED DESCRIPTION:
Zambia has high rates of women of childbearing age infected with Human Immune Deficiency Virus (HIV). The majority (93%) engage in intravaginal practices (here referred to as IVP) by internal cleansing (intravaginal cleansing) or by inserting products inside the vagina (intravaginal insertion). IVP are culturally driven practices associated with an increased risk of HIV transmission and may play an important role in exacerbating the HIV epidemic across sub-Saharan Africa.

This application proposes to 1) evaluate the long term impact of a bio-behavioral intervention targeting VP among HIV infected women (n=128) in Lusaka, Zambia, and 2) assess the relative contributions of VP and bacterial vaginosis (BV) to lower genital tract inflammation and HIV shedding. Study aims will address the following:

Aim 1. To develop and evaluate the long term impact of a culturally tailored bio-behavioral intervention aimed to decrease IVP in HIV positive women and evaluate the relative contribution of IVP and BV to lower genital inflammation and shedding of HIV.

Aim 1.1. To develop and evaluate the long term impact of a bio-behavioral intervention to decrease IVP.

Intra vaginal practices, as culturally driven and condoned behaviors, are difficult to modify. It is hypothesized that a culturally tailored bio-behavioral intervention is needed to decrease IVP, and that women participating in the intervention condition will reduce IVP in comparison with women in a time matched control condition. Experimental approach: Women engaging in IVP will be randomly assigned to one of two conditions (intervention or control). IVP will be evaluated and compared over 12 months.

Aim 1.2. To compare rates of BV, lower genital tract inflammatory markers and HIV shedding in HIV infected women engaging in VP with and without BV.

Due to the close relationship between IVP and BV, it is difficult to determine the relative contribution of each to lower genital tract inflammation and HIV shedding. It is hypothesized that women engaging in IVP with BV will have similar levels of both lower genital tract inflammatory cytokines and HIV viral load to those without BV. Experimental approach: Vaginal secretions and cervicovaginal fluid will be collected from women engaging in IVP. The presence of BV, inflammatory cytokines (IL-6 and IL-8), and HIV RNA will be determined by gram stain, ELISA and PCR techniques respectively, and compared in women that engage in IVP with and without BV.

Aim 1.3. To compare BV, lower genital inflammatory markers and shedding of HIV in HIV seropositive women participating in the intervention versus control condition.

Interventions to decrease IVP have the goal of reducing BV and associated adverse health outcomes. It is hypothesized that the bio-behavioral intervention will decrease BV, lower genital tract inflammation and HIV shedding. Experimental approach: Laboratory assessments used for Aim 1.2 will be repeated and compared at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women recruited
* Living with HIV-1 infection
* At least 18 years of age,
* Receiving antiretroviral therapy
* Intravaginal practices
* Vaginal intercourse with men in the month prior to enrolment
* Living in the Lusaka metropolitan area

Exclusion Criteria:

* Pregnant
* Being on hormonal contraception
* Having an intrauterine device (IUD) in place to avoid the potential for induced changes in inflammatory cytokines in the genital mucosa due to contraception.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants were women living with HIV-1 infection, at least 18 years of age, receiving antiretroviral therapy (ART), engaging in intravaginal practices and vaginal intercourse with men in the month prior to enrolment, and living in the Lusaka metropolitan area. Because the primary outcomes were intravaginal practices and bacterial vaginosis, participants had to be female.
Enrollment: 128 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2014-02-05 (Actual); Study Completion 2014-02-05 (Actual)

PRIMARY OUTCOMES:
Vaginal Practices | 12-months
  Information on intravaginal practices was collected using a culturally tailored questionnaire assessing specific products used for IVP. Questions to assess product use in the prior month utilized a dichotomous response option: product use (1 = yes, 0 = no).

CONTACTS AND LOCATIONS:
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Available from the PI upon request.

REFERENCES:
- [Background] Alcaide ML, Chisembele M, Mumbi M, Malupande E, Jones D. Examining targets for HIV prevention: intravaginal practices in Urban Lusaka, Zambia. AIDS Patient Care STDS. 2014 Mar;28(3):121-7. doi: 10.1089/apc.2013.0309. Epub 2014 Feb 25. PMID 24568672
- [Background] Alcaide ML, Chisembele M, Malupande E, Arheart K, Fischl M, Jones DL. A cross-sectional study of bacterial vaginosis, intravaginal practices and HIV genital shedding; implications for HIV transmission and women's health. BMJ Open. 2015 Nov 9;5(11):e009036. doi: 10.1136/bmjopen-2015-009036. PMID 26553833
- [Background] Alcaide ML, Cook R, Chisembele M, Malupande E, Jones DL. Determinants of intravaginal practices among HIV-infected women in Zambia using conjoint analysis. Int J STD AIDS. 2016 May;27(6):453-61. doi: 10.1177/0956462415585447. Epub 2015 May 8. PMID 25957322
- [Derived] Alcaide ML, Chisembele M, Malupande E, Rodriguez VJ, Fischl MA, Arheart K, Jones DL. A bio-behavioral intervention to decrease intravaginal practices and bacterial vaginosis among HIV infected Zambian women, a randomized pilot study. BMC Infect Dis. 2017 May 12;17(1):338. doi: 10.1186/s12879-017-2436-3. PMID 28494795